CLINICAL TRIAL: NCT00092365
Title: A Randomized, Placebo-Controlled, Parallel-Group, Double -Blind Study to Evaluate the Safety and Efficacy of Rofecoxib 12.5 mg and Celecoxib 200 mg in Patients With Osteoarthritis of the Knee
Brief Title: A Study of Two Approved Drugs in Patients With Osteoarthritis (0966-220)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0966-220; 2004_071
Record Dates: First submitted 2004-09-22; First posted 2004-09-27 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — rofecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0966, rofecoxib
Drug: Comparator: celecoxib, placebo

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of two approved drugs in the treatment of osteoarthritis of the knee.

DETAILED DESCRIPTION:
The duration of treatment is 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee which requires treatment with medication for pain relief

Exclusion Criteria:

* Any known allergy to the study drugs

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2003-04-01 (Actual); Primary Completion 2003-11-01 (Actual); Study Completion 2003-11-01 (Actual)

PRIMARY OUTCOMES:
Osteoarthritis (OA) of the knee as measured by Patient Global Assessment of Response to Therapy (PGART) and WOMAC VA 3.0 over 6 weeks of treatment.

SECONDARY OUTCOMES:
OA of the knee as measured by PGART over 6 wks of treatment.
WOMAC Question #1 over 6 wks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Birbara C, Ruoff G, Sheldon E, Valenzuela C, Rodgers A, Petruschke RA, Chang DJ, Tershakovec AM. Efficacy and safety of rofecoxib 12.5 mg and celecoxib 200 mg in two similarly designed osteoarthritis studies. Curr Med Res Opin. 2006 Jan;22(1):199-210. doi: 10.1185/030079906X80242. PMID 16393445
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html